CLINICAL TRIAL: NCT04832152
Title: Testing the Feasibility of a Teletherapy Plus Parent Coaching Intervention for Children With Autism
Brief Title: Telehealth Intervention for Autism Spectrum Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 412579-19406
Record Dates: First submitted 2021-03-24; First posted 2021-04-05 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: The purpose of this project is to adapt an existing, evidence-based occupational therapy intervention for children with ASD to a telehealth delivery model. The main objectives of the project are to 1) adapt the manual so that it operationalizes best-practices of occupational therapy telehealth50,51, 2) test its feasibility, and 3) evaluate preliminary outcomes.
  Design: In the formative research aspect of this project will use survey methodology and a modified Delphi process to adapt our current intervention to a telehealth delivery model (Aim 1).
  In Aim 2 we will conduct a feasibility trial (Figure 2) to assess therapists' fidelity, participant recruitment and retention, acceptability of the protocol by parents and therapists, and clinically meaningful differences.
Masking Description: none. This is a feasiblity trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility trial group (Other): One group (arm) trial where all will receive treatment.
  Interventions: Other: OT4ASD

INTERVENTIONS:
Other: OT4ASD — Occupational therapy will focus on education and coaching of families/caregivers of children with autism spectrum disorder to help them adapt their daily routines to address their child's sensory needs.

SUMMARY:
Autism Spectrum Disorder (ASD) is one of the most frequently occurring childhood-onset neurodevelopmental disorders affecting 1 in every 54 children. Most children with ASD experience challenges participating in daily activities (e.g.: eating, sleeping, bathing, grooming, playing, etc.) and receive occupational therapy intervention to address these. The COVID-19 pandemic has restricted in-person therapy for many of these children and there is an urgent need for evidence-based, validated telehealth intervention. This project will adapt an evidence-based occupational therapy intervention, termed OT4ASD to a telehealth delivery model. The aims of the project are to: 1) adapt the existing intervention protocol to a telehealth delivery model, 2) train therapists and evaluate the therapist's ability to conduct OT4ASD, 3) determine if OT4ASD delivered via the telehealth is acceptable and feasible to parents and interventionists; and 4) whether children improve in the daily living skills. OT4ASD follows a systematic protocol and uses active, individually-tailored sensory motor activities that are specifically designed to address the child's needs. The investigators believe this will be the first telehealth manualized protocol to address the sensory motor symptoms of ASD and measure outcomes at the daily life activity and participation levels.

DETAILED DESCRIPTION:
Autism Spectrum Disorder (ASD) is one of the most frequently occurring childhood-onset neurodevelopmental disorders affecting 1 in every 54 children1. As a lifelong condition, individuals with ASD experience a range of intellectual, behavioral, sensory, motor, and functional challenges that impact successful participation in daily life activities and tasks. As a result, occupational therapy (OT) intervention is a frequently requested and utilized service in ASD, and clinically validated OT approaches are needed. In a series of studies funded by the NIH and autism foundations, our team manualized and studied an OT intervention that targets the sensory and motor factors impacting participation in daily life activities and tasks and showed significant improvements in those that received the intervention in comparison to controls 2-4. In this project, the investigators plan to adapt our existing protocol to a telehealth model of service delivery, and evaluate its feasibility and preliminary effectiveness.

The COVID-19 global pandemic created a call to action for healthcare providers to design unique and innovative methods for therapeutic service delivery. This shift creates an urgent need for remote solutions so that therapeutic services can be delivered in safely and effectively. Since the onset of the COVID-19 pandemic, families have reported regression in adaptive functioning in addition to a negative impact on social skills and increased anxiety, and an impact to daily routines of children with ASD5. In a recent survey of families with children with ASD, 95% of the parents reported that disruptions in services/therapies negatively impacted their child's behaviors and only 35% of families were receiving telehealth services/therapies6. To address these increased needs for children with ASD and to meet the need of manualized telehealth intervention, the investigators propose to adapt the existing intervention to a telehealth delivery model. This intervention, termed occupational therapy for children with Autism Spectrum Disorder (OT4ASD) targets the sensory motor factors that impact behavior and participation in life activities and tasks. This project is significant in that it will address the need for evidence-based OT services for children with ASD using an innovative telehealth model. Given that many children with ASD require treatment for the sensory and motor symptoms that impact their optimal participation in a range of daily life activities and tasks, and that the current COVID 19 pandemic has compromised access to this therapy, this project is urgently needed.

Innovation: Telehealth offers an emerging and innovative approach for OT intervention. Research shows that children with ASD require intensive intervention to assure best outcomes and telehealth offers an innovative solution for providing therapy during a pandemic. To the investigator's knowledge, this will be the first telehealth manualized protocol to address the sensory motor symptoms of ASD and measure outcomes at the activity and participation levels of the ICF framework. Importantly, the investigators will adapt an evidence-based, manualized intervention with solid data on outcomes to a telehealth model. The protocol will operationalize the data-driven decision making (DDDM) approach into an on-line format. DDDM is innovative in that it explicitly guides the therapist to contextualize intervention within the child and family's real life participation challenges and use data from assessment to individualize the intervention. DDDM measures outcomes at the proximal (sensory and motor factors) and distal (functional/participation-based goals) levels facilitating an intervention that is context-specific and participation-oriented.

Methods: The project will first adapt the existing protocol into a telehealth delivery model using a formative approach that includes a modified Delphi process to obtain input and consensus from experts in telehealth and autism interventions and key stakeholders (parents and clinical interventionists). Next, the investigators will conduct a feasibility trial to assess the acceptability, satisfaction and implementation fidelity as well as gather data on clinically meaningful outcomes. Outcomes will be measured at the proximal and distal levels using validated outcome measures to assure information gained is relevant and scientifically rigorous. Data from the feasibility trial will be used to support an R01 application to conduct a randomized trial of OT4ASD.

To implement the project, the investigators utilize a highly skilled team of clinicians and scientists with experience in conducting randomized trials in autism who will work collaboratively to translate knowledge gained into useful information that will impact the lives of families and children with ASD. Our approach is consistent with contemporary models of evidence-based practice and rehabilitation science promoting promote high integrity, evidence-based information from research that targets relevant and meaningful areas for each child and family. The timeline is ambitious and the investigators feel well-equipped to meet it given past experiences and expertise.

In summary, this project addresses an urgent need to provide rehabilitation services to children with ASD using remote technology. It will operationalize best practices in telehealth to adapt an existing evidence-based OT intervention and utilize a skilled and experienced team of investigators. As such, this project is consistent with the AACPDM mission to promote excellence in research and services for persons with childhood-onset disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism Spectrum Disorder
* Between the ages of 4 years 0 months and 12 years 0 months
* Evidence of sensory symptoms based on the Sensory Processing Measure
* Family is willing to participate
* Physically able to participate in active, sensorimotor activities

Exclusion Criteria:

* Primary (visual or auditory) uncorrected sensory deficits
* Do not meet age or diagnostic criteria

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Daily Living Skills Change Score - Pediatric Evaluation of Disabilities Inventory | up to 14 weeks
  Change in daily living skills (on a scale of 0 to 25) measured with the Pediatric Evaluation of Disabilities Inventory. Change score range 0-25; higher score means better outcome.
Pervasive Developmental Disorders Behavioral Inventory T Score Autism Behaviors | up to 14 weeks
  Change is autism behaviors and sensory approach behaviors. Raw scores are converted to T Score. Minimum = 10 Maximum = 80

SECONDARY OUTCOMES:
Goal Attainment Scale T Score | up to 14 weeks
  Rating of individual goals. Rating Scale -2 to +2 is converted to T-Score; higher score means better outcome.
Sensory Processing Measure | up to 14 weeks
  Change in sensory hypo or hyper reactivity. T scores range from 40 to 80; Lower score means better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Rose R. Kennedy Children's Evaluation and Rehabilitation Center (CERC) at Montefiore, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Publication in high impact autism journal, and presentation at international autism research meetings.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available following completion of the study and publication of findings.
Access Criteria: Upon written request (reviewed by principal investigator) information will be shared.